CLINICAL TRIAL: NCT01524536
Title: Assessment of Glucocorticoid Responsiveness and Mechanisms of Resistance in Hypereosinophilic Syndromes
Brief Title: Steroid Treatment for Hypereosinophilic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120026; 12-I-0026
Record Dates: First submitted 2012-02-01; First posted 2012-02-02 (Estimated); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-02-22

CONDITIONS: Eosinophilia; Hypereosinophilic Syndrome; Leukocyte Disorder; Hematologic Diseases
Keywords: Hypereosinophilia; Hypereosinophilic Syndrome; Corticosteroids; Therapy; HES
MeSH Terms: conditions — Eosinophilia; Hypereosinophilic Syndrome; Leukocyte Disorders; Hematologic Diseases | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Steroid Challenge (Other): A single oral dose of prednisone (1 mg/kg rounded to the nearest 5mg) was administered to all participants. The following day, participant began glucocorticoid therapy of prednisone 30 mg oral daily for one week followed by a standardized taper until a minimally effective dose was achieved or participant tapered to prednisone 5 mg oral daily.
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: prednisone — Glucocorticoids (GC) are considered the first- line therapy for hypereosinophilic syndrome.

SUMMARY:
Background:

- Hypereosinophilic syndrome (HES) is a disorder in which the body has too many eosinophils (a type of white blood cell). Too many eosinophils in HES can cause damage to the heart, nerves, or skin. Certain drugs can help lower eosinophil counts to prevent tissue damage. Corticosteroids, such as prednisone, are used for initial therapy in this disorder. Although most people respond to prednisone, some people develop side effects from it, or do not respond very well to treatment. Better ways of determining the dose to give could help to decide on the best therapy for HES.

Objectives:

* To determine whether a single-dose of prednisone can be used to predict which people with hypereosinophilia respond to treatment.
* To study lack of response to steroid treatment in people with HES.

Eligibility:

Inclusion criteria:

* Individuals with hypereosinophilic syndrome with high eosinophil counts.
* Individuals who are willing to have blood drawn before and after getting steroids.

Exclusion criteria:

* Individuals who are on more than 10mg of prednisone (or similar drug)
* Individuals with hypereosinophilic syndrome who are on other medications that could interfere with the study
* Women who are pregnant or breast-feeding
* Individuals who have a known gene mutation associated with chronic eosinophilic leukemia
* Children less than 18 years old who weigh less than 48kg or 106lb

Design:

* Participants will have a screening visit with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will have a single dose of the steroid prednisone by mouth in the morning. Blood samples will be collected 2, 4, 24 hours after this dose.
* On the day after the steroid dose, participants will provide another blood sample in the morning.
* Participants will start to take prednisone daily when they return home. Blood samples will be collected weekly at the participant s doctor s office. The dose of prednisone will be lowered depending on the weekly eosinophil count. We will try to get each person on the lowest dose of prednisone possible that will control the disorder. Participants who do not respond or have severe side effects will be taken off prednisone. Other treatments will be considered for people who do not respond to steroids. The goal is to evaluate the response to prednisone. Our research will try to figure out why some people do not respond to steroids. Most people will complete the study within 6 to 16 weeks, depending on their response to prednisone.

DETAILED DESCRIPTION:
This study aims to develop a model to determine whether a single, oral, weight-based dose of glucocorticoid (GC) can predict clinical and biologic response to GC s over the long term in subjects with hypereosinophilic syndrome (HES). Subjects with FIP1L1/PDGFRalpha-negative HES, who are symptomatic with eosinophil count >1500/microL and receiving less than or equal to10 mg prednisone daily, will be enrolled. A single oral dose of prednisone (1 mg/kg rounded to the nearest 5mg) will be administered. Eosinophil count and various laboratory parameters will be assessed at 2 hours, 4 hours and 24 hours following prednisone administration (investigators will be blinded to the results of the eosinophil counts). The subjects will then begin GC therapy at 30 mg prednisone daily followed by a standardized taper. The lowest dose of GC at which symptoms and eosinophilia are controlled will be compared to the change in eosinophil count at 2, 4 and 24 hours post-challenge. Mechanisms and in vitro correlates of GC resistance will also be explored.

ELIGIBILITY:
* SUBJECT INCLUSION CRITERIA:

Subjects on Protocol #94-I-0079 will be eligible for participation in the study only if all of the following criteria apply:

1. Subjects must be 7 years of age or older to enroll
2. Subject meets diagnostic criteria for HES (AEC >1500/microL, absence of a secondary cause and signs and/or symptoms attributable to the eosinophilia)
3. AEC greater than 1500 microL obtained within 14 days prior to enrollment
4. Willingness to perform the timed steroid challenge
5. Appropriate candidate for GC treatment after challenge
6. Willingness to have samples stored for future research

SUBJECT EXCLUSION CRITERIA:

A subject will not be eligible to participate in the study if any of the following apply:

1. Receiving >10 mg prednisone or equivalent at the time of enrollment.
2. Receiving less than or equal to 10 mg of prednisone or equivalent but have not been on a fixed dose for at least 3 weeks (subjects on a current corticosteroid taper will be excluded).
3. AEC less than or equal to 1500/microl on the day of the steroid challenge
4. Use of immunomodulatory medications, (other than less than or equal to 10 mg/day prednisone) including but not limited to biologics, within the past 6 months.
5. Pregnant at the time of screening.
6. Have a known mutation in the FIP1L1-PDGFR gene.
7. Any condition that, in the opinion of the investigator, places the subject at undue risk by participating in the protocol.
8. Weight less than 48 kg (106 lbs) in subjects less than 18 years of age.

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-02-16 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paneez Khoury, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ogbogu PU, Bochner BS, Butterfield JH, Gleich GJ, Huss-Marp J, Kahn JE, Leiferman KM, Nutman TB, Pfab F, Ring J, Rothenberg ME, Roufosse F, Sajous MH, Sheikh J, Simon D, Simon HU, Stein ML, Wardlaw A, Weller PF, Klion AD. Hypereosinophilic syndrome: a multicenter, retrospective analysis of clinical characteristics and response to therapy. J Allergy Clin Immunol. 2009 Dec;124(6):1319-25.e3. doi: 10.1016/j.jaci.2009.09.022. PMID 19910029
- [Background] Prin L, Lefebvre P, Gruart V, Capron M, Storme L, Formstecher P, Loiseau S, Capron A. Heterogeneity of human eosinophil glucocorticoid receptor expression in hypereosinophilic patients: absence of detectable receptor correlates with resistance to corticotherapy. Clin Exp Immunol. 1989 Dec;78(3):383-9. PMID 2612051
- [Background] Hamilos DL, Leung DY, Muro S, Kahn AM, Hamilos SS, Thawley SE, Hamid QA. GRbeta expression in nasal polyp inflammatory cells and its relationship to the anti-inflammatory effects of intranasal fluticasone. J Allergy Clin Immunol. 2001 Jul;108(1):59-68. doi: 10.1067/mai.2001.116428. PMID 11447383
- [Derived] Stokes K, Yoon P, Makiya M, Gebreegziabher M, Holland-Thomas N, Ware J, Wetzler L, Khoury P, Klion AD. Mechanisms of glucocorticoid resistance in hypereosinophilic syndromes. Clin Exp Allergy. 2019 Dec;49(12):1598-1604. doi: 10.1111/cea.13509. Epub 2019 Oct 27. PMID 31657082
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-I-0026.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 participants were consented to protocol but three did not meet the eligibility criteria so did not start study.
Period: Overall Study
Arm/Group | Steroid Challenge
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Steroid Challenge
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 1
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Eosinophil Count After Glucocorticoid Challenge
Description: Response to glucocorticoid challenge as assessed by the percentage of the eosinophil count 24 hours post-glucocorticoid challenge relative to the Baseline AEC for each participant.
  Measure Description (%): Percent of baseline AEC is defined as the Absolute Eosinophil Count at 24 hours divided by the Absolute Eosinophil Count at Baseline *100.
Time Frame: 24 hours
Population: All participants who received the single challenge dose of prednisone
Measure: Mean (95% Confidence Interval); unit: percentage of eosinophil count
Groups:
- Steroid Challenge - Responders; Steroid Challenge - Non-responders: A single oral dose of prednisone (1 mg/kg rounded to the nearest 5mg) was administered to all participants. The following day, participant began glucocorticoid therapy of prednisone 30 mg oral daily for one week followed by a standardized taper until a minimally effective dose was achieved or participant tapered to prednisone 5 mg oral daily.
Arm/Group | Steroid Challenge - Responders | Steroid Challenge - Non-responders
Number analyzed (Participants) | 16 | 7
percentage of eosinophil count | -69.6 [-80.1 to -59.1] | -13.6 [-35.2 to 9.13]

2. Secondary Outcome: Participants With Glucocorticoid Responsiveness - IHES Variant
Description: Participants with idiopathic hypereosinophilic syndromes (IHES) that achieved glucocorticoid responsiveness, suboptimal responsiveness, or without response.
Time Frame: Baseline (Day 1)
Population: All participants who received the prednisone challenge and completed dose course post challenge
Measure: Count of Participants; unit: Participants
Groups:
- Steroid Challenge - Glucocorticoid Responsiveness: Participants with hypereosinophilic syndromes (IHES) that achieved glucocorticoid responsiveness defined as final minimally effective dose of prednisone of 0mg-15mg
- Steroid Challenge - Glucocorticoid Suboptimal Responsiveness: Participants with hypereosinophilic syndromes (HES) with suboptimal glucocorticoid responsiveness defined as achieving final minimally effective dose of prednisone of 16mg-40mg
- Steroid Challenge - Glucocorticoid Unresponsiveness: Participants with hypereosinophilic syndromes (HES) that were not responsive to prednisone defined as no decline of absolute eosinophil count (AEC) below 1000/mm^3 after one week of prednisone 30 mg daily, followed by 2 days of prednisone 60 mg daily
Arm/Group | Steroid Challenge - Glucocorticoid Responsiveness | Steroid Challenge - Glucocorticoid Suboptimal Responsiveness | Steroid Challenge - Glucocorticoid Unresponsiveness
Number analyzed (Participants) | 11 | 5 | 7
Participants | 6 | 2 | 2

3. Secondary Outcome: Participants With Glucocorticoid Responsiveness - LHES Variant
Description: Participants with lymphoid hypereosinophilic syndromes (LHES) that achieved glucocorticoid responsiveness, suboptimal responsiveness, or without response.
Time Frame: Baseline (Day 1)
Population: All participants who received the prednisone challenge and completed dose course post challenge
Measure: Count of Participants; unit: Participants
Groups:
- Steroid Challenge - Glucocorticoid Responsiveness: Participants with hypereosinophilic syndromes (HES) that achieved glucocorticoid responsiveness defined as final minimally effective dose of prednisone of 0mg-15mg
Arm/Group | Steroid Challenge - Glucocorticoid Responsiveness | Steroid Challenge - Glucocorticoid Suboptimal Responsiveness | Steroid Challenge - Glucocorticoid Unresponsiveness
Number analyzed (Participants) | 11 | 5 | 7
Participants | 2 | 1 | 2

4. Secondary Outcome: Participants With Glucocorticoid Responsiveness - MHES Variant
Description: Participants with myeloid hypereosinophilic syndromes (MHES) that achieved glucocorticoid responsiveness, suboptimal responsiveness, or without response.
Time Frame: Baseline (Day 1)
Population: All participants who received the prednisone challenge and completed dose course post challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Challenge - Glucocorticoid Responsiveness | Steroid Challenge - Glucocorticoid Suboptimal Responsiveness | Steroid Challenge - Glucocorticoid Unresponsiveness
Number analyzed (Participants) | 11 | 5 | 7
Participants | 0 | 0 | 1

5. Secondary Outcome: Participants With Glucocorticoid Responsiveness - Overlap HES Subtypes
Description: Participants with overlap hypereosinophilic syndromes that achieved glucocorticoid responsiveness, suboptimal responsiveness, or without response.
Time Frame: Baseline (Day 1)
Population: All participants who received the prednisone challenge and completed dose course post challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Challenge - Glucocorticoid Responsiveness | Steroid Challenge - Glucocorticoid Suboptimal Responsiveness | Steroid Challenge - Glucocorticoid Unresponsiveness
Number analyzed (Participants) | 11 | 5 | 7
Participants | 3 | 2 | 1

6. Secondary Outcome: Mean Baseline IgE Level
Description: Mean baseline immunoglobulin E (IgE) level in participants prior to initiation of glucocorticoid
Time Frame: Baseline (Day 1)
Population: All participants who received the prednisone challenge and completed dose course post challenge
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Steroid Challenge - Glucocorticoid Responsiveness | Steroid Challenge - Glucocorticoid Suboptimal Responsiveness | Steroid Challenge - Glucocorticoid Unresponsiveness
Number analyzed (Participants) | 11 | 5 | 7
IU/mL | 285.2 [50.74 to 1603] | 1171.5 [69.23 to 19824] | 434.8 [27.49 to 6877]

7. Secondary Outcome: Mean Baseline Absolute Eosinophil Count
Description: Mean baseline absolute eosinophil count in participants prior to initiation of glucocorticoids
Time Frame: Baseline (Day 1)
Population: All participants who received the prednisone challenge and completed dose course post challenge
Measure: Geometric Mean (95% Confidence Interval); unit: 10^3 cells per microliter
Arm/Group | Steroid Challenge - Glucocorticoid Responsiveness | Steroid Challenge - Glucocorticoid Suboptimal Responsiveness | Steroid Challenge - Glucocorticoid Unresponsiveness
Number analyzed (Participants) | 11 | 5 | 7
10^3 cells per microliter | 2.81 [2.097 to 3.771] | 3.85 [2.036 to 7.313] | 5.90 [2.772 to 12.59]

8. Secondary Outcome: Participants With Glucocorticoid Responsiveness - Cardiac Involvement
Description: Cardiac involvement in participants with hypereosinophilic syndromes (HES)
Time Frame: Baseline (Day 1)
Population: All participants who received the prednisone challenge and completed dose course post challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Challenge - Glucocorticoid Responsiveness | Steroid Challenge - Glucocorticoid Suboptimal Responsiveness | Steroid Challenge - Glucocorticoid Unresponsiveness
Number analyzed (Participants) | 11 | 5 | 7
Participants | 1 | 0 | 4

9. Secondary Outcome: Participants With Glucocorticoid Responsiveness - Pulmonary Involvement
Description: Pulmonary involvement in participants with hypereosinophilic syndromes (HES)
Time Frame: Baseline (Day 1)
Population: All participants who received the prednisone challenge and completed dose course post challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Challenge - Glucocorticoid Responsiveness | Steroid Challenge - Glucocorticoid Suboptimal Responsiveness | Steroid Challenge - Glucocorticoid Unresponsiveness
Number analyzed (Participants) | 11 | 5 | 7
Participants | 4 | 3 | 3

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Steroid Challenge
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 7/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Steroid Challenge (N=23)
Glaucoma (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Swelling face (General disorders) | 1
Thirst (General disorders) | 1
Weight increased (Investigations) | 2
Fluid retention (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT01524536/Prot_SAP_000.pdf